CLINICAL TRIAL: NCT05652673
Title: Safe Stop IPI-NIVO Trial: Early Discontinuation of Nivolumab Upon Achieving a (confirmed) Complete or Partial Response in Patients with Irresectable Stage III or Metastatic Melanoma Treated with First-line Ipilimumab-nivolumab
Brief Title: Safe Stop Ipilimumab-nivolumab (IPI-NIVO) Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, A.A.M. van der Veldt, Doctor, Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL82177.078.22
Record Dates: First submitted 2022-08-12; First posted 2022-12-15 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Melanoma Stage IV; Melanoma Stage III; Immunotherapy; Toxicity, Drug
MeSH Terms: conditions — Melanoma; Drug-Related Side Effects and Adverse Reactions | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Early discontinuation of nivolumab (Experimental)
  Interventions: Drug: nivolumab

INTERVENTIONS:
Drug: nivolumab — Early discontinuation of nivolumab maintenance therapy in patients with irresectable stage III or metastatic melanoma

SUMMARY:
Safe Stop IPI-NIVO Trial: Early discontinuation of nivolumab upon achieving a (confirmed) complete or partial response in patients with irresectable stage III or metastatic melanoma treated with first-line ipilimumab-nivolumab

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Irresectable stage III or metastatic melanoma
* Treated with at least one dose of first-line ipilimumab-nivolumab and considered to be a candidate for maintenance treatment with nivolumab:

  * previous systemic treatment, including immune-checkpoint inhibitors, in (neo)adjuvant setting for resectable melanoma is allowed
  * in this protocol, nivolumab maintenance is interchangeable with pembrolizumab maintenance therapy.
* Response evaluation according to RECIST v1.1 30 using a diagnostic CT documenting target lesions every 12 (-2/+6) weeks from the start of ipilimumab-nivolumab:

  * for patients with CR on a diagnostic CT at response evaluation, a low-dose CT (which is usually part of 18FDG-PET/CT) is allowed at baseline
  * for patients with PR on a diagnostic CT at response evaluation, a low-dose CT (which is usually part of 18FDG-PET/CT) is allowed if sufficient target lesions are measurable for response evaluation according to RECIST v1.1 criteria 30
  * in case of asymptomatic brain metastases prior to start of first-line ipilimumab-nivolumab, intracerebral tumor response should be confirmed using an MRI for response evaluation prior to inclusion in this study.
* Patients should be included after first CR/PR or first confirmed CR/PR according to RECIST v1.1 30:

  * inclusion should take place no later than 5 weeks after first confirmed CR/PR
  * in case of SD at first response evaluation, confirmed CR/PR is required for inclusion
  * planned and willing to discontinue nivolumab within 4(+1) weeks after inclusion, i.e. first CR/PR or first confirmed CR/PR
  * no later than 9 months after start of treatment with ipilimumab-nivolumab
* Presence of MRI brain for the screening of brain metastases (prior to discontinuation of ipilimumab-nivolumab)
* Participants with previously locally treated brain metastases may participate in case they meet the following criteria:

  * completely asymptomatic brain metastases at inclusion
  * MRI of brain at baseline and for response evaluation during treatment
* Signed and dated informed consent form

Exclusion Criteria:

* Patients with SD/PD according to RECIST v1.1
* Malignant disease other than being treated in this study. Exceptions to this exclusion include the following: malignancies that were treated curatively and have not recurred within 2 years prior to start of study treatment; completely resected basal cell and squamous cell skin cancers and any completely resected carcinoma in situ.
* Presence of symptomatic brain metastases:

  * prior to first-line treatment with ipilimumab-nivolumab, or;
  * when defined as new or progressive brain metastases at the time of study entry;
  * brain metastases with need for steroid treatment in the last 8 weeks prior to study entry Note: An incidental epileptic seizure caused by a brain lesion is not considered an exclusion criterion.

(provided that the other in- and exclusion criteria are met);

* Presence of leptomeningeal metastases;
* Systemic chronic steroid therapy (>10mg/day prednisone or equivalent) at inclusion or patients who need or needed any other second-line immunosuppressive therapy (e.g. infliximab, mycophenolate mofetil) for the treatment of immune related adverse events (irAEs). Note: local steroids such as topical, inhaled, nasal and ophthalmic steroids are allowed.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Ongoing response | 12 months after start of ipilimumab-nivolumab combination therapy
  The rate of ongoing response at 12 months in patients with irresectable stage III or metastatic melanoma who are treated with first-line ipilimumab-nivolumab and who early discontinue nivolumab upon achieving a CR or PR according to RECIST v1.1

SECONDARY OUTCOMES:
Ongoing response | 24 months after start of treatment
  Ongoing response at 24 months after start of first-line treatment with ipilimumab-nivolumab
Disease control | 5 years after inclusion
  Disease control (CR/PR) at different time points
duration of response | 5 years after inclusion
  Duration of response (CR/PR) measured until progressive/recurrent disease
Melanoma Specific Survival rate | 5 years after inclusion
  Melanoma specific survival measured from start of first-line treatment with ipilimumab-nivolumab until melanoma related death
Overall Survival | 5 years after inclusion
  Overall survival (OS) measured from start of first-line treatment with ipilimumab-nivolumab until death by any cause
(serious) adverse events | 5 years after inclusion
  Impact of discontinuation treatment on (S)AEs
ORR | 5 years after inclusion
  Overall Response Rate (ORR) per RECIST v1.1 in retreated patients
Re-treatment | 5 years after inclusion
  Rate of re-treatment for melanoma
Disease control (CR/PR/SD [stable disease]/not PD [progressive disease]) after restarting (systemic) treatment for melanoma | 5 years after inclusion
  Disease control (CR/PR/SD [stable disease]/not PD [progressive disease]) after restarting (systemic) treatment for melanoma
Quality of life questionnaires EuroQoL EQ-5D-5 | 5 years after inclusion
  Quality of life is measured using questionnaires: EuroQoL EQ-5D-5

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Janssen JC, van Dijk B, de Joode K, Aarts MJB, van den Berkmortel FWPJ, Blank CU, Boers-Sonderen MJ, van den Eertwegh AJM, de Groot JWB, Jalving M, de Jonge MJA, Joosse A, Kapiteijn E, Kamphuis-Huismans AM, Naipal KAT, Piersma D, Rikhof B, Westgeest HM, Vreugdenhil G, Oomen-de Hoop E, Mulder EEAP, van der Veldt AAM. Safe Stop IPI-NIVO trial: early discontinuation of nivolumab upon achieving a complete or partial response in patients with irresectable stage III or metastatic melanoma treated with first-line ipilimumab-nivolumab - study protocol. BMC Cancer. 2024 May 23;24(1):632. doi: 10.1186/s12885-024-12336-0. PMID 38783238